CLINICAL TRIAL: NCT04367740
Title: ScreenNC: A Study to Determine the Number of Asymptomatic Individuals Who Have Antibodies to the SARS-CoV-2 Infection
Brief Title: ScreenNC, a Study to Determine the Number of Asymptomatic Individuals Who Have Antibodies to the Virus That Causes COVID-19
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0937
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-01

CONDITIONS: Asymptomatic Condition; Infection Viral; Coronavirus Infections; Severe Acute Respiratory Syndrome Coronavirus 2; Coronaviridae Infections; RNA Virus Infections; Virus Diseases; Communicable Disease
Keywords: COVID-19; Pandemic; COVID-19 virus testing
MeSH Terms: conditions — Asymptomatic Diseases; Virus Diseases; Coronavirus Infections; Coronaviridae Infections; RNA Virus Infections; Communicable Diseases; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood; virus from nasal or oral swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Serum Antibodies: Blood samples to be obtained assess for IgG antibodies against SARS-CoV2
  Interventions: Diagnostic Test: To assess for development of IgG antibodies against SARS-CoV2

INTERVENTIONS:
Diagnostic Test: To assess for development of IgG antibodies against SARS-CoV2 — Swabs will be collected to assess for COVID-19 if PPE supplies allow.
  Other Names: Nasopharyngeal Swab; Oropharyngeal Swab

SUMMARY:
Purpose: To determine the number of asymptomatic individuals who have antibodies to SARS-CoV-2, the virus which causes COVID-19

DETAILED DESCRIPTION:
ScreenNC is design ed for comprehensive virus screening and serology to assess exposure to SAR-CoV2 in persons not-indicated for COVID-19 testing as per the CDC screening algorithm and implemented at UNC Health Care (at the time of activation). This trial is designed to generate point prevalence of infected (I) persons, independent of clinical symptoms. The susceptible (S) class is the number of COVID-19 tested by any FDA-approved NP swab test or a SARS-CoV2 IgG antibody test. At present FDA does not have approved SARS-CoV serology and such serology is not used for diagnosis of acute infection. The recovered (R) class is the number of positives. This information allows for modeling of the COVID-19 epidemic in NC. The investigation is not testing the effectiveness or safety of either of these testing modalities, though serology may be offered in the future by UNC Healthcare laboratories. The blood samples to be obtained assess development of host response to SARS-CoV2 infection.

ScreenNC will be implemented within the logistic and clinical limitations of the current outbreak. This is a single visit study. Since there is a shortage of PPE the investigators will rely on screening at locations different then the screening of presumed infected persons. Additionally, due to logistical considerations, volunteers may have a viral swab (nasopharyngeal or oropharyngeal) and/or a blood sample obtained. Thus, at recruitment, volunteers may be asked to give both samples or only one.

Viral load testing will be done at LabCorp and/or UNC labs using compatible assays (Roche, ThermoFischer , WHO). Confirmatory testing (other PCR, sequencing, culture) will be done at UNC. Blood samples will be tested at the McClendon Clinical Immunology laboratory for IgG antibodies against SARS-CoV2.

Because these patients are in the UNC Health Care system, The investigators will have access to their medical records, which will provide very granular information as to co-morbidities and other demographic factors which can be assessed in the context of SAR-CoV-2 (COVID-19) infection status. Future analyses of this cohort will employ statistical methods which allow us to account for sampling bias of this convenience sample to construct a representative sample of the state of NC .

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-99 who arrive at any participating UNC Healthcare clinic for care and who have a medical record in UNC EPIC.
* Patients may be included if they have completed the quarantine as recommended by the CDC and at least 4 weeks since the initial positive COVID-19 NP test.

Exclusion Criteria:

* Any individual arriving at any participating UNC Healthcare clinic for diagnosis or treatment of respiratory symptoms meeting the following COVID-19 clinical evaluation criteria:

  1. Developed non-allergy respiratory symptoms of cough or shortness of breath in the past 7 days

     AND
  2. Meet ONE OR MORE of these criteria

     * Had close contact (within 6 feet for 10 or more minutes) with a person diagnosed with COVID-19
     * Works in a healthcare setting
     * Is pregnant or postpartum within 2 weeks of delivery
     * Is morbidly obese: BMI = 40 or 100 pounds over ideal body weight
     * Diabetes mellitus
     * Immunosuppression, including caused by medications or by HIV infection
     * Pulmonary disease, including asthma
     * Cardiovascular disease
     * Hypertensive disease
     * Renal disease
     * Hepatic disease
     * Hematologic disease, including sickle cell disease
     * Neurological condition that limits movement
     * Moderate to severe developmental delay

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients seen at UNC Outpatient clinics who are asymptomatic for COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 6313 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Asymptomatic patients with an IgG response from SARS-CoV-2 infection. | at enrollment
  Presence or absence of IgG antibodies to SARS-CoV2

SECONDARY OUTCOMES:
Percentage of Asymptomatic patients with viral presence of SARS-CoV-2 infection. | at enrollment
  swab for presence of SARS-CoV-2 virus

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No